CLINICAL TRIAL: NCT06280677
Title: An Observational Study to Evaluate the Expression Profiles of Oocyte-potency-related Genes in Cumulus Cells of Women Treated With Human Recombinant FSH (Hr-FSH)and Triggered With GnRH Agonist in an Oocyte Donation Program
Brief Title: Aurora Test for ART Donor Patients (AURORA-Donor)
Status: Recruiting | Type: Observational
Sponsor: Fertiga, Belgium (Industry)
Collaborators: Fertilab (Unknown); Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023.Aurora-Donor
Record Dates: First submitted 2024-01-31; First posted 2024-02-28 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GnRH Antagonist & hr-FSH: Patients stimulated with GnRH Antagonist & hr-FSH with GnRH Agonist trigger
  Interventions: Other: AURORA-Donor
- Progesterone & hr-FSH: Patients stimulated with Progesterone & hr-FSH with GnRH Agonist trigger
  Interventions: Other: AURORA-Donor

INTERVENTIONS:
Other: AURORA-Donor — Explorative study of cumulus cells gene expression in relation to the oocyte competence for good quality blastocyst formation and predictive for clinical pregnancy.

SUMMARY:
This is a randomized observational study. The main aim is to determine potential oocyte competence predictive mRNA expression profiles in the cumulus cells isolated form individual oocytes. In 2 patient cohorts: 1)GnRH Antagonist & hr-FSH with GnRH Agonist trigger, 2) Progesterone & hr-FSH with GnRH Agonist trigger.

ELIGIBILITY:
Inclusion Criteria Donor:

* Patients are 18 to 35 years old
* BMI between 17-30
* Regular menstrual cycles
* AFC > 8
* Patient profile in compliance with SEF (Sociedad Española de Fertilidad) directives for egg donation (medical, psychological and genetic screening, informed consent)
* Patients' stimulation: GnRH Antagonist & hr-FSH with GnRH Agonist trigger or Progesterone & hr-FSH with GnRH Agonist trigger
* Patients agree that the oocytes will be denuded for cumulus testing and provide written informed consent for participation to the study

Exclusion Criteria Donor:

* BMI < 17 or > 30
* Extreme irregular menstrual cycles (<20 days or >40 days)
* AFC < 8
* <8 MII on previous egg retrieval
* Women with history of poor oocyte maturation or known maturation defect or unexplained failure in previous treatments
* Patients that fail to comply with SEF (Sociedad Española de Fertilidad) directives for egg donation (medical, psychological and genetic screening, informed consent)

Inclusion Criteria Recipient:

* Patients applying for ART egg donation with fresh/frozen sperm from the partner or frozen donor sperm. With eSB-FET in modified natural cycle or an HRT cycle.
* Patients are from 18 to 50 years old.
* Patients will be treated by ICSI (intracytoplasmic sperm injection) and eSB-FET (elective Single Blastocyst Frozen Embryo Transfer)
* Recipient patients agree that the donors' oocytes will be denuded for cumulus testing and provide written informed consent for participation to the study

Exclusion Criteria for oocyte Recipients

* Patient included in any other prospective study.
* BMI < 17 or > 35
* Severe uterine factor: Multiple myomectomy, multiple fibroids, major uterine malformation (unicorn, septum), Asherman Sd, severe adenomyosis
* Repeated Implantation Failure or Repeated Pregnancy Loss after euploid Single Blastocyst Transfer
* Severe male factor: Abnormal Caryotype or FISH, severe OAT / Cripto-Azoospermia, DNA Fragmentation >50% after medical treatment
* TESE / TESA (testicular sperm extraction/aspiration)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Donor's for this study must be between 18 and 35 years of age, and compliant with SEF directive for egg donation. Only patient with at least 6 MII will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Basic clinical donor patient and stimulation characteristics: P4 | During ovarian stimulation (max 3 weeks)
  Serum values for P4 (ng/ml)
Basic clinical donor patient and stimulation characteristics: E2 | During ovarian stimulation (max 3 weeks)
  Serum values for E2 (ng/L)
Basic clinical donor patient and stimulation characteristics: Gonadotropin type and dose | During ovarian stimulation (max 3 weeks)
  Gonadotropin type and dose (IU) used for stimulation
Clinical evaluation: number of Follicles | During ovarian stimulation (max 3 weeks)
  The number of follicles at time of trigger (oocyte-pick-up day-2)
Clinical evaluation: number of cumulus-oocyte complex | Day 1 of embryo culture
  The number of cumulus-oocyte complex at time of pick-up
Clinical evaluation: Meiosis II oocytes | Day 1 of embryo culture
  The number of meiosis II oocytes (nominator) divided by the total number of oocytes retrieved (denominator)
Clinical evaluation: Abnormal fertilization | Day 1 of embryo culture
  The number of abnormal fertilized oocytes on day 1 at 17+1h post insemination, as a function of all COC's inseminated
Clinical evaluation: Normal Fertilization | Day 1 of embryo culture
  The number of fertilized oocytes on day 1 (presence of 2PN and 2PB assessed at 17 + 1h post-insemination), as a function of all COC's inseminate
Clinical evaluation: Day 3 embryo evaluation | Day 3 of embryo culture
  Day 3 embryo morphology evaluation according to the standard of care of the ART clinic
Clinical evaluation: Day 5/6 embryo evaluation | Day 6 of embryo culture
  Day 5/6 embryo evaluation based on the criteria of Gardner and Schoolcraft (Gardner and Schoolcraft 1999)
Clinical evaluation: Day5/6 good quality blastocyst rate | Day 6 of embryo culture
  Defined as the proportion of 2PN zygotes which are good-quality blastocyst on Day 5/6 (116 +-2h and 140 +-2h post-insemination) (ESHRE Special Interest Group of Embryology and Alpha Scientists in Reproductive Medicine 2017)
Clinical evaluation: Embryo utilization | Day 6 of embryo culture
  Defined as the number of blastocyst suitable for cryopreservation and transfer as a function of the number of normally fertilized (2PN) oocytes observed on day 1 (ESHRE Special Interest Group Alpha Scientists 2017)
Expression profile: blastocyst formation | 2.5 years after study start
  The expression profiles of cumulus of oocyte leading to a blastocyst and the expression profiles of cumulus of oocyte not leading to a blastocyst has been determined using RNA-Seq.

SECONDARY OUTCOMES:
Biochemical pregnancy | Day 10 after embryo transfer
  A pregnancy diagnosed only by the detection of beta human chorionic gonadotropin (hCG) in serum or urine
Clinical pregnancy with positive fetal heartbeat | week 5-6 after embryo transfer
  Pregnancy diagnosed by ultrasonographic or clinical documentation of at least one fetus with a discernible heartbeat in gestational week 6 to 8
Expression profile: pregnancy prediction | 2.5 years after study start
  The expression profile of cumulus of oocytes leading to pregnancy and the expression profiles of oocytes not leading to pregnancy are established using RNA seq.
Normalized messenger ribonucleic acid (mRNA) expression | 2.5 years after study start
  Quantitative Polymerase Chain Reaction (QPCR) data of samples informative for blastocyst formation and pregnancy prediction have been collected

OTHER OUTCOMES:
Ongoing pregnancy rate | Week 10-11 after embryo transfer
  The presence of gestational sacs with fetal heart beat detected by transvaginal ultrasound examination in gestational week 10 to 11
Live birth | week 24-42 after embryo transfer
  is defined as the birth of at least one newborn after 24 weeks gestation that exhibits any sign of live (twins will be a single count)
Cumulative pregnancy | 2.5 years after study start
  The accumulated ongoing pregnancy after fresh and frozen-warmed embryo transfers within one stimulation cycle. Pregnancy with detectable heart rate at ≥ 12 weeks gestation after the completion of the first transfer.
  Live birth is defined as the birth of at least one newborn after 24 weeks gestation that exhibits any sign of live (twins will be a single count)
Cumulative live birth | 2.5 years after study start
  The number of deliveries with at least one live birth resulting from one initiated or aspirated ART cycle, including all cycles in which fresh and/or frozen embryos are transferred, until one delivery with a live birth occurs or until all embryos are used, whichever occurs first.
Miscarriage rate | week 22 after embryo transfer
  the spontaneous loss of an intra-uterine pregnancy prior to 22 completed weeks of gestational age

CONTACTS AND LOCATIONS:
Locations (1):
- Fertilab, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No